CLINICAL TRIAL: NCT05117385
Title: The Effect of the Consumption of 4 Botanical Extracts (Acerola, Panax Ginseng, Echinacea, Quillaja) on the Innate and Adaptive Immune Response in Healthy Adults: a Pilot Randomized Placebo-controlled Clinical Trial
Brief Title: The Effect of the Consumption of 4 Botanical Extracts on Immunity in Healthy Adults (B-4-Immune)
Acronym: B-4-Immune
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-A01973-38
Record Dates: First submitted 2021-11-10; First posted 2021-11-11 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Healthy Subject; Immunity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Acerola (Experimental): dietary supplement : acerola extract self administrated by mouth for 28 days
  1 capsule per day
  Interventions: Dietary Supplement: Botanical extract
- Panax ginseng extract (Experimental): dietary supplement : panax ginseng extract self administrated by mouth for 28 days
  1 capsule per day
  Interventions: Dietary Supplement: Botanical extract
- Echinacea extract (Experimental): dietary supplement : echinacea extract self administrated by mouth for 28 days
  1 capsule per day
  Interventions: Dietary Supplement: Botanical extract
- Quillaja extract (Experimental): dietary supplement : quillaja extract self administrated by mouth for 28 days
  1 capsule per day
  Interventions: Dietary Supplement: Botanical extract
- Maltodextrin (Placebo Comparator): dietary supplement : maltodextrin supplement self administrated by mouth for 28 days
  1 capsule per day
  Interventions: Dietary Supplement: Botanical extract

INTERVENTIONS:
Dietary Supplement: Botanical extract — 1 capsule per day

SUMMARY:
This study will evaluate the capacity of botanical extracts to modulate immune mechanisms compared to a placebo group in healthy volunteers.

DETAILED DESCRIPTION:
In this ex-vivo pilot study, healthy volunteers will consume extracts during 28 days and blood will be sampled at baseline and end of study. The purpose of this study is to evaluate the ex vivo immune responses with and without stimulation after consumption of botanical extracts and identify the main mechanisms involved. The effect of the consumption of 4 botanical extracts on the quality of life in healthy adults compared to placebo will be also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60 years (limits included)
* 18,5 < Body Mass Index < 30 kg/m2
* Without modification of their normal eating/drinking habits, body weight and physical activity patterns in the last 4 weeks
* Consumption of citrus fruits and fruit juices limited to two servings per day maximum in the last 7 days
* Consumption of caffeine < 400 mg/day in the last 2 weeks
* For non-menopausal women: with the same reliable contraception (oral or local hormonal contraception, surgery (ligation, bilateral ovariectomy), copper intrauterine device) since at least 3 cycles before the beginning of the study and agreeing to keep it during the entire duration of the study
* For menopausal women: without hormone replacement therapy
* Daily consumption of alcohol less than 2 glasses
* Non-smoking or tobacco consumption stopped for at least 12 months
* Good general and mental health according to the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form
* Affiliated with a social security scheme
* Accepts to be registered to the VRB site (Volunteers in Biomedical Research database)

After V0 biological analysis the subjects will be eligible to the study on the following criteria:

* Normal values of complete blood count (CBC), hemoglobin, hematocrit, MVC (mean corpuscular volume), MCH (mean corpuscular haemoglobin), HCT (haematocrit), MCHC mean corpuscular haemoglobin concentration), RDW (Red cells Distribution width), MPV (mean platelet volume), PCT (plateletcrit), ASAT (aspartate aminotransferase), ALAT (alanine aminotransferase), urea, creatinine, HDL-cholesterol, LDL-cholesterol, total cholesterol, TG (triglycerides), glycemia according to the investigators' opinion
* Negative pregnancy test: blood beta HCG < 5 IU/L for women in childbearing age

Exclusion Criteria:

* Any vaccination 6 weeks before inclusion visit and/or any vaccination during the study
* Specific food diet/habits: high protein or vegan diet
* Subjects who exercise more than 150 min per weeks of intense activity (which ask for an important physical effort and need to breathe much more than usual; for example, lift heavy load, mountain biking, playing football..) and more than 5 hours per week of moderate activity (which ask for a moderate physical effort and need to breathe a little bit more than usual; for example lift moderate load, quiet biking… )
* With a past or current allergic rhinitis (sneezing, eye and nose scratching) and/or asthma (cough, wheezing, shortness of breath)
* With a current or past disorder of neuropathy / diabetic neuropathy
* Suffering from a metabolic or endocrine disorder
* SBP > 139 and/or DBP > 89 mmHg
* Treated or untreated diabetes and/or any pancreatic disease
* With a current or past cardiac disease
* With a current or past liver disease (cirrhosis, fibrosis, NASH…)
* With a current or past pulmonary disease
* With a current or past renal disease
* With a significant risk of bladder/kidney stones
* Infectious disease in the last 6 weeks
* Untreated hypo/hyperthyroidism, or uncontrolled hypo/hyperthyroidism or treated hypo/hyperthyroidism for less than 3 months (treated hypo/hyperthyroidism stabilized for at least 3 months is accepted)
* Untreated hypertension, or uncontrolled hypertension, or treated hypertension for less than 3 months (treated hypertension stabilized for at least 3 months is accepted)
* Untreated hypercholesterolemia or uncontrolled hypercholesterolemia or treated hypercholesterolemia for less than 3 months according to the investigator's opinion (treated and controlled hypercholesterolemia stabilized for at least 3 months is accepted according to the investigator's opinion)
* Past or current inflammatory disease with an impact on immune responses (rheumatoid arthritis, bone metabolic disease, psoriasis, gout, symptomatic chondrocalcinosis and active infection…)
* Immunodeficient volunteer and/or current immunosuppressive therapy
* With a current or past auto-immune disease or immunodeficiency
* Gastrointestinal disease, gastroenteritis (within 4 weeks), intestinal occlusion, prolonged severe diarrhea, severe regurgitation, difficulty for swallowing
* Current cancer or in remission < 5 years and/or any past or current hematological cancers (exception: basal cell carcinoma, or non-squamous cell skin cancer, prostate cancer, or in situ carcinoma without any significative progression in the past 2 years)
* Antibiotics consumption in the past 3 months
* Chronic antiviral and/or antibacterial treatment
* Current heparin treatment or anti-coagulation drug
* Consumption of laxative in the past 3 months
* Subjects who take, nasal steroids, decongestants, antihistamines, combination cold formulas, anti-inflammatory drugs (nonsteroidal anti-inflammatory drugs, ibuprofen, cyclo-oxygenase 2 inhibitors) and therapy with immunostimulants (cytokines, thymus fractions) in the last 4 weeks
* Consumption of any food supplement (including but not limited to omega-3-fatty acid, probiotic supplements, vitamin, mineral supplement, herbal immunostimulant, etc…) in the last 4 weeks
* Bariatric surgery or any disease that could lead to intestinal malabsorption of the study products
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient
* Pregnant and/or breastfeeding women or intending to become pregnant in the next 3 months
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator
* Currently participating to another clinical trial or volunteer who has ended his participation to a previous clinical study in the past 90 days
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision
* Presenting a psychological or linguistic incapability to sign the informed consent
* Impossible to contact in case of emergency

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-07-18 (Estimated); Study Completion 2022-07-18 (Estimated)

PRIMARY OUTCOMES:
Ex vivo Immune blood cell response after challenges at baseline (before supplementation) and after 28 days of each botanical consumption compared to placebo | 28 days
  Innate immunity like response and adaptative cell activation

SECONDARY OUTCOMES:
1. Frequency of innate and adaptative immune cell before and after 28 days of consumption of each botanical extract compared to placebo | 28 days
  The variation between both visits of the frequency of several circulating cells from innate and adaptative immunity expressed in % of white blood cells and absolute values
2. Variation of quality of life before and after 28 days of consumption of each botanical extract compared to placebo | 28 days
  Assessed by the SF-12-v2 (Short-Form Health Survey version 2) questionnaire. it is a generic patient-reported measure of health status that provides summary scores of physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Krausz, PhD, Study Director — Givaudan France Naturals
Locations (1):
- Biofortis Merieux Nutrisciences, Saint-Herblain, France